CLINICAL TRIAL: NCT06278701
Title: Effects of Late-evening Snacks on Nutritional Status and Metabolic Pattern of Patients With Primary Hepatocellular Carcinoma After Hepatectomy
Brief Title: The Effect of Late-evening Snacks on Patients With Primary Hepatocellular Carcinoma After Hepatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DU Yao (Other)
Responsible Party: Sponsor-Investigator, DU Yao, Pharmacist-in-charge, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-003-01
Record Dates: First submitted 2024-02-05; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Liver Neoplasms
Keywords: Liver cancer; late evening snack; Metabolic pattern; Nutritional status
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This study utilizes a grouping method based on patient preference. You will learn about the 2 dietary modalities, the late-evening snacks and the regular diet, and then you will be placed in the different groups according to your preference. Patients who volunteer for the 1h bedtime meal will be in the test group and those who volunteer for the regular diet will be in the control group. Dietary counseling and follow-up visits will be conducted in both groups, the difference being the presence or absence of the 1h bedtime meal pattern.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (No Intervention): Patients who voluntarily accept a regular diet and do not eat again 1h before bedtime
- the test group (Experimental): Patients who voluntarily accepted to have an additional meal 1h before bedtime (total calories 200-275kcal, protein 11.5g-18g, complex carbohydrates 25-55g).
  Interventions: Other: late-evening snacks

INTERVENTIONS:
Other: late-evening snacks — have an additional meal 1h before bedtime (total calories 200-275kcal, protein 11.5g-18g, complex carbohydrates 25-55g).
  Arms: the test group

SUMMARY:
Late-evening snacks, in which a portion of food is moved to bedtime while the total amount of food eaten per day remains unchanged, can effectively improve the metabolic state of accelerated catabolism.

The goal of this clinical trial is to learn about the effects of late-evening snacks on health conditions of hepatocellular carcinoma patients who underwent hepatectomy, and to further explore the effects of late-evening snacks on patients' metabolic patterns. The main question it aims to answer are: • the effect of late-evening snacks on the nutritional status of hepatic resection patients with hepatocellular carcinoma;

* the effect of late-evening snacks on the recovery of liver function in liver cancer hepatectomy patients;
* the effect of late-evening snacks on the complication rate of hepatic resection patients with hepatocellular carcinoma;
* the effect of late-evening snacks on long-term quality of life of hepatic resection patients with hepatocellular carcinoma;
* the effect of late-evening snacks on the metabolic pattern of hepatic resection patients with hepatocellular carcinoma.

After learning about the 2 dietary modalities of the late-evening snacks and regular diet, patients will be placed in the different groups according to your preference. Patients who enter the test group will have additional meal 1h before bedtime every day, while patients in the control group will have normal diet. Patients will be asked to :

* eat 1h before bedtime;
* follow the doctor's instructions during their stay in the hospital;
* have follow-up examinations at 1 month, 3 months and 6 months after the operation, after which blood samples will be collected for metabolite testing.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years;
* Meet the diagnostic criteria of China's "Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2022 Edition)", clinically diagnosed with primary liver cancer, hospitalized with radical hepatectomy as the main surgical treatment, no indication of metastasis of the tumor to extra-hepatic organs in preoperative tests and examinations, no absolute contraindications to surgery, complete resection of the liver tumor in the operation, and hepatocellular carcinoma confirmed by postoperative pathological diagnosis；
* Child-Pugh grades A and B;
* Preoperative Eastern Cooperative Oncology Group Physical Status Score (ECOG-PS) of 0 to 2;
* The patient is conscious, has normal verbal communication, and is able to cooperate with the relevant examinations;
* Fully informed about the study and voluntarily signed an informed consent form.

Exclusion Criteria:

* Failure to meet selection criteria;
* Nutritional assessment as cachexia;
* Presence of contraindications to enteral nutrition (EN) or EN intolerance, such as acute gastrointestinal bleeding, intestinal obstruction.(≥ grade 3, National Cancer Institute-Common Terminology Criteria for Adverse Events [NCINCI-CTCAE v 5.0]);
* Simultaneous combination of malignant tumors in other parts of the body;
* Combined hepatic encephalopathy or definite infection on admission;
* Known refractory metabolic diseases (e.g., poorly controlled diabetes mellitus or fasting glucose ≥10 mmol/L, hyperthyroidism, hypothyroidism, metabolic acidosis)；
* Decreased renal function (defined as serum creatinine Cr level ≥176.8 μmol/L);
* Intravenous or oral nutritional supplements, such as proteins, amino acids, etc., applied within one month prior to admission to the hospital;
* Patients with severe stress or severe complications such as respiratory failure with severe cardiac, hepatic, renal and other insufficiencies；
* Persons with mental and neurological disorders who are unable to cooperate with a physician;
* Alzheimer's disease, cerebral atrophy, acute stage or sequelae of cerebrovascular disease, cognitive impairment;
* Previously poor adherence to medication and nutritional counseling;
* Critically ill and difficult to assess;
* On the liver transplant waiting list or under consideration for liver transplantation, as such patients may discontinue follow-up before the end of the study;
* Less than 12 months since last localized treatment (TACE or HAIC or ablative therapy);
* Other circumstances that the researcher considers inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Albumin rising | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum albumin levels in patients at each time point

SECONDARY OUTCOMES:
Prealbumin rising | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum levels of prealbumin in patients at each time point
Decrease in Alanine Aminotransferase | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum levels of alanine aminotransferase in patients at each time point
Decrease in Aspartate Aminotransferase | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum levels of aspartate aminotransferase in patients at each time point
Decrease in Cholinesterase | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum levels of cholinesterase in patients at each time point
Decrease in Total bilirubin | Day 1 of admission/Post-operative day 6/1 month postoperative/3 months postoperative/6 months postoperative
  Serum levels of total bilirubin in patients at each time point
Lower total hospitalization costs | From admission to discharge，an average of 1 month
  Total cost from patient hospitalization to discharge
Relapse-Free Survival | From the time the patient underwent hepatectomy until the date of first recording to the date of progression or death from any cause, whichever comes first, assessed up to 2 years
  Time from when the patient achieved complete remission after hepatectomy to the time of recurrence or cutoff for follow-up
Improved quality of life | 1 month postoperative/3 months postoperative/6 months postoperative
  Patients completed EORTC QLQ-C30 at various time points

CONTACTS AND LOCATIONS:
Overall Officials: Yao Du, Master, Study Director — Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Tsilimigras DI, Bagante F, Sahara K, Moris D, Hyer JM, Wu L, Ratti F, Marques HP, Soubrane O, Paredes AZ, Lam V, Poultsides GA, Popescu I, Alexandrescu S, Martel G, Workneh A, Guglielmi A, Hugh T, Aldrighetti L, Endo I, Pawlik TM. Prognosis After Resection of Barcelona Clinic Liver Cancer (BCLC) Stage 0, A, and B Hepatocellular Carcinoma: A Comprehensive Assessment of the Current BCLC Classification. Ann Surg Oncol. 2019 Oct;26(11):3693-3700. doi: 10.1245/s10434-019-07580-9. Epub 2019 Jul 2. PMID 31267302
- [Background] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739
- [Background] Liu PH, Hsu CY, Hsia CY, Lee YH, Huang YH, Chiou YY, Lin HC, Huo TI. Surgical Resection Versus Radiofrequency Ablation for Single Hepatocellular Carcinoma </= 2 cm in a Propensity Score Model. Ann Surg. 2016 Mar;263(3):538-45. doi: 10.1097/SLA.0000000000001178. PMID 25775062
- [Background] Borhofen SM, Gerner C, Lehmann J, Fimmers R, Gortzen J, Hey B, Geiser F, Strassburg CP, Trebicka J. The Royal Free Hospital-Nutritional Prioritizing Tool Is an Independent Predictor of Deterioration of Liver Function and Survival in Cirrhosis. Dig Dis Sci. 2016 Jun;61(6):1735-43. doi: 10.1007/s10620-015-4015-z. Epub 2016 Jan 2. PMID 26725059
- [Background] Rong W, Xia H, Zhang K, Zhang Y, Tao C, Wu F, Wang L, Zhang H, Sun G, Wu J. Serum metabolic effects of corn oligopeptides with 7-day supplementation on early post-surgery primary liver cancer patients: a double-blind randomized controlled trial. Hepatobiliary Surg Nutr. 2022 Dec;11(6):834-847. doi: 10.21037/hbsn-21-116. PMID 36523946
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale RG, Waitzberg D, Bischoff SC, Singer P. ESPEN practical guideline: Clinical nutrition in surgery. Clin Nutr. 2021 Jul;40(7):4745-4761. doi: 10.1016/j.clnu.2021.03.031. Epub 2021 Apr 19. PMID 34242915
- [Result] Huang TH, Hsieh CC, Kuo LM, Chang CC, Chen CH, Chi CC, Liu CH. Malnutrition associated with an increased risk of postoperative complications following hepatectomy in patients with hepatocellular carcinoma. HPB (Oxford). 2019 Sep;21(9):1150-1155. doi: 10.1016/j.hpb.2019.01.003. Epub 2019 Feb 11. PMID 30765200
- [Result] Puri P, Dhiman RK, Taneja S, Tandon P, Merli M, Anand AC, Arora A, Acharya SK, Benjamin J, Chawla YK, Dadhich S, Duseja A, Eapan CE, Goel A, Kalra N, Kapoor D, Kumar A, Madan K, Nagral A, Pandey G, Rao PN, Saigal S, Saraf N, Saraswat VA, Saraya A, Sarin SK, Sharma P, Shalimar, Shukla A, Sidhu SS, Singh N, Singh SP, Srivastava A, Wadhawan M. Nutrition in Chronic Liver Disease: Consensus Statement of the Indian National Association for Study of the Liver. J Clin Exp Hepatol. 2021 Jan-Feb;11(1):97-143. doi: 10.1016/j.jceh.2020.09.003. Epub 2020 Oct 1. PMID 33679050
- [Result] Joliat GR, Kobayashi K, Hasegawa K, Thomson JE, Padbury R, Scott M, Brustia R, Scatton O, Tran Cao HS, Vauthey JN, Dincler S, Clavien PA, Wigmore SJ, Demartines N, Melloul E. Guidelines for Perioperative Care for Liver Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations 2022. World J Surg. 2023 Jan;47(1):11-34. doi: 10.1007/s00268-022-06732-5. Epub 2022 Oct 30. PMID 36310325
- [Result] Plauth M, Bernal W, Dasarathy S, Merli M, Plank LD, Schutz T, Bischoff SC. ESPEN guideline on clinical nutrition in liver disease. Clin Nutr. 2019 Apr;38(2):485-521. doi: 10.1016/j.clnu.2018.12.022. Epub 2019 Jan 16. PMID 30712783
- [Result] Amodio P, Bemeur C, Butterworth R, Cordoba J, Kato A, Montagnese S, Uribe M, Vilstrup H, Morgan MY. The nutritional management of hepatic encephalopathy in patients with cirrhosis: International Society for Hepatic Encephalopathy and Nitrogen Metabolism Consensus. Hepatology. 2013 Jul;58(1):325-36. doi: 10.1002/hep.26370. Epub 2013 May 31. PMID 23471642
- [Result] Leoni L, Valoriani F, Barbieri R, Pambianco M, Vinciguerra M, Sicuro C, Colecchia A, Menozzi R, Ravaioli F. Unlocking the Power of Late-Evening Snacks: Practical Ready-to-Prescribe Chart Menu for Patients with Cirrhosis. Nutrients. 2023 Aug 5;15(15):3471. doi: 10.3390/nu15153471. PMID 37571408
- [Result] Guo YJ, Tian ZB, Jiang N, Ding XL, Mao T, Jing X. Effects of Late Evening Snack on Cirrhotic Patients: A Systematic Review and Meta-Analysis. Gastroenterol Res Pract. 2018 Apr 1;2018:9189062. doi: 10.1155/2018/9189062. eCollection 2018. PMID 29805447
- [Result] Chen CJ, Wang LC, Kuo HT, Fang YC, Lee HF. Significant effects of late evening snack on liver functions in patients with liver cirrhosis: A meta-analysis of randomized controlled trials. J Gastroenterol Hepatol. 2019 Jul;34(7):1143-1152. doi: 10.1111/jgh.14665. Epub 2019 May 7. PMID 30883904
- [Result] Nakaya Y, Okita K, Suzuki K, Moriwaki H, Kato A, Miwa Y, Shiraishi K, Okuda H, Onji M, Kanazawa H, Tsubouchi H, Kato S, Kaito M, Watanabe A, Habu D, Ito S, Ishikawa T, Kawamura N, Arakawa Y; Hepatic Nutritional Therapy (HNT) Study Group. BCAA-enriched snack improves nutritional state of cirrhosis. Nutrition. 2007 Feb;23(2):113-20. doi: 10.1016/j.nut.2006.10.008. PMID 17234504
- [Result] Takeshita S, Ichikawa T, Nakao K, Miyaaki H, Shibata H, Matsuzaki T, Muraoka T, Honda T, Otani M, Akiyama M, Miuma S, Ozawa E, Fujimito M, Eguchi K. A snack enriched with oral branched-chain amino acids prevents a fall in albumin in patients with liver cirrhosis undergoing chemoembolization for hepatocellular carcinoma. Nutr Res. 2009 Feb;29(2):89-93. doi: 10.1016/j.nutres.2008.12.005. PMID 19285598
- [Result] Harima Y, Yamasaki T, Hamabe S, Saeki I, Okita K, Terai S, Sakaida I. Effect of a late evening snack using branched-chain amino acid-enriched nutrients in patients undergoing hepatic arterial infusion chemotherapy for advanced hepatocellular carcinoma. Hepatol Res. 2010 Jun;40(6):574-84. doi: 10.1111/j.1872-034X.2010.00665.x. PMID 20618455
- [Result] Morihara D, Iwata K, Hanano T, Kunimoto H, Kuno S, Fukunaga A, Yotsumoto K, Takata K, Tanaka T, Sakurai K, Iwashita H, Ueda S, Hirano G, Yokoyama K, Nakane H, Nishizawa S, Yoshikane M, Anan A, Takeyama Y, Kakumitsu S, Kitamura Y, Sakamoto M, Irie M, Shakado S, Sohda T, Watanabe H, Sakisaka S. Late-evening snack with branched-chain amino acids improves liver function after radiofrequency ablation for hepatocellular carcinoma. Hepatol Res. 2012 Jul;42(7):658-67. doi: 10.1111/j.1872-034X.2012.00969.x. Epub 2012 Mar 2. PMID 22380706
- [Result] Tripodi F, Badone B, Vescovi M, Milanesi R, Nonnis S, Maffioli E, Bonanomi M, Gaglio D, Tedeschi G, Coccetti P. Methionine Supplementation Affects Metabolism and Reduces Tumor Aggressiveness in Liver Cancer Cells. Cells. 2020 Nov 16;9(11):2491. doi: 10.3390/cells9112491. PMID 33207837
- [Result] Koreeda C, Seki T, Okazaki K, Ha-Kawa SK, Sawada S. Effects of late evening snack including branched-chain amino acid on the function of hepatic parenchymal cells in patients with liver cirrhosis. Hepatol Res. 2011 May;41(5):417-22. doi: 10.1111/j.1872-034X.2011.00795.x. PMID 21518402

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT06278701/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT06278701/ICF_001.pdf